CLINICAL TRIAL: NCT05651386
Title: The Six Food Elimination in Postprandial Distress Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s63494
Record Dates: First submitted 2020-02-12; First posted 2022-12-15 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Six food elimination diet (Other): The six food elimination diet will be performed in all subjects.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — No blinded, no controlled intervention.

SUMMARY:
The six food elimination diet, as known in eosinophilic esophagitis, will be performed in 15 patients with functional dyspepsia (subtype postprandial distress syndrome). Screening will exclude patients with allergies by performing immunocaps on blood. Before and after the 8 weeks of diet, an gastroduodenoscopy with biopsies will be performed to evaluate duodenal eosinophilia, mast cells and permeability. To evaluate gastric sensorimotor function, a gastric emptying breath test and a barostat test will be performed before and after the diet.

Symptoms will be monitored with a daily diary (LPDS diary) and food intake will be evaluated during 2 weeks.

If there is an improvement of symptoms during the diet, a reintroduction period will start. This period will last 6 weeks. Every 2 weeks, two food groups will be reintroduced. When there is a clear worsening in symptoms, a new endoscopy with biopsies will be performed.

DETAILED DESCRIPTION:
To assess the effect of the six food elimination diet on duodenal eosinophilia, an interventional study will be conducted in 15 patients.

The study design includes 8 weeks of a strict 6 food elimination diet, followed by an 8 week reintroduction phase in patients with symptom improvement. The duration of 8 weeks is based on the effect of the 6 FED in eosinophilic esophagitis.

Each subject will undergo a screening before the start of the diet. During the screening visit, all study procedures will be explained, the informed consent form will be signed by the participant, and the inclusion and exclusion criteria will be checked by revising the participant's medical history and by using screening GI symptom questionnaires (Rome IV questionnaire).

The screening visit will include a physical examination, medical history and a blood sample for IgE testing to exclude typical food allergies.

When eligibility is confirmed during the screening visit, a fourteen-day period starts. In this period, the LPDS diary (Leuven Postprandial distress syndrome) and food diary will be filled out on a daily basis to assess symptoms at baseline. The food diary will be available via an application for mobile phones or online use. The Comprehensive Nutrition Assessment Questionnaire will be filled in to analyse baseline food intake.

At visit 1, following tests will be conducted in a 2-day period (outpatient clinic):

* A gastroduodenoscopy with biopsies, optionally/preferably under sedation.
* A gastric barostat study.
* A gastric emptying breath test. If desired, the gastric emptying test can be performed at home and sent or taken to the clinic.
* Questionnaires (as specified in chapter 10.3.) After these tests, the 6 food elimination diet (6FED) will be explained by a trained dietician.

The diet will be followed during 8 weeks under supervision of this dietician with experience in eosinophilic esophagitis.

During the 6FED the compliance of patients will be evaluated by the use of diet diaries from week 6 to 8. Symptoms will be evaluated throughout the 8-week dietary restriction period using the daily LPDS diary. Patients will report daily food intake via an application for mobile phone or online use during two weeks of the diet period.

A telephone call will be scheduled after two and six weeks, to assess compliance.

After 8 weeks of six food elimination diet, a new gastroduodenoscopy with biopsies will be performed, as well as a new gastric barostat and gastric emptying breath test, as described at visit 1.

At visit 2, patients with a symptom improvement, defined as an average LPDS with 0.5 point or more compared to baseline will be sent for a consultation with our dietician for the explanation of reintroduction of nuts and fish.

This will be done in a non-blinded way.

During the reintroduction period, patients will visit the hospital every 2 weeks for visit 3, 4 and 5. First, fish and nuts will be reintroduced, than eggs and soy and lastly gluten and milk. Patients with symptom worsening, defined as an average LPDS with 0.5 point or more compared to the end of the 6FED diet period, will be invited to undergo a with gastroscopy with biopsies and a new blood sample for PBMCs.

During the entire study, patients will fill in the daily diary (LPDS).

ELIGIBILITY:
Inclusion Criteria:

* Functional dyspepsia patients with meal related symptoms (Rome IV Postprandial Distress Syndrome, PDS)
* Witnessed written informed consent prior to any study procedures
* Patients aged between 18 and 70 years inclusive
* Male or female patients
* Women of child-bearing potential agree to apply a highly effective method of birth control during the entire duration of the trial. Women of non-childbearing potential may be included if surgically sterile or postmenopausal with at least 2 year without spontaneous menses.
* Subject is capable to understand the study and the questionnaires, and to comply with the study requirements.

Exclusion Criteria:

* History of gastrointestinal surgery (other than appendectomy).
* Organic gastro-intestinal disease
* Major psychiatric disorder
* Patients with eosinophilic esophagitis
* Presence of diabetes mellitus
* Presence of coeliac disease, lupus, scleroderma and other systemic auto-immune disease.
* Active H. Pylori infection or < 6 months after eradication
* Predominant irritable bowel syndrome (IBS)
* Predominant gastro-oesophageal reflux disease (GERD)
* Atopic constitution or food allergy
* Ongoing diet which interferes with the 6 food elimination diet.
* Drugs altering gastric emptying or anti-inflammatory drugs
* Females who are pregnant or lactating
* Patients not capable to understand or be compliant with the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-02-19 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Duodenal eosinophilia | 8 weeks
  Measured with duodenal biopsies with H&E staining

SECONDARY OUTCOMES:
Duodenal mast cells | 8 weeks
  Measured with duodenal biopsies with immunohistochemistry
Duodenal permeability | 8 weeks
  Measured with duodenal biopsies with ussing chambers
PDS symptoms | 8 weeks
  Measured with daily symptom diary (LPDS)
Functional dyspepsia symptoms | 8 weeks
  Measured with PAGI-SYM
Symptom severity | 8 weeks
  Measured with OSS
Overall symptom improvement | 8 weeks
  Measured with OTE
Quality of life | 8 weeks
  Measured with SF-NDI

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, PhD, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No